CLINICAL TRIAL: NCT02098486
Title: Antibiotic Prophylaxis for ERCP: a Comparison of Intravenous Ceftriaxone With Intravenous Moxifloxacin in the Prophylaxis of Cholangitis
Brief Title: Comparisons of Intravenous Ceftriaxone With Intravenous Moxifloxacin in ERCP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Hong Joo Kim, Associate Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERCPMOXIVSCEF
Record Dates: First submitted 2014-03-22; First posted 2014-03-28 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Cholangitis
Keywords: Bile duct obstruction; Cholangitis; Moxifloxacin; Ceftriaxone; Sepsis
MeSH Terms: conditions — Cholangitis; Cholestasis; Sepsis | interventions — Moxifloxacin; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftraxone (Active Comparator): ceftriaxone (2 g/day, diluted in 40 cc of 5% dextrose water, infused more than 30 min)
  Interventions: Drug: ceftriaxone
- Moxifloxacin (Active Comparator): Intravenous moxifloxacin (400 mg/day, infused more than 60 min)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin
  Arms: Moxifloxacin
Drug: ceftriaxone
  Arms: Ceftraxone

SUMMARY:
Background and aims: The use of prophylactic antibiotics before endoscopic retrograde cholangiopancreatography (ERCP) is recommended by all major international gastroenterological societies, especially in the presence of an obstructed biliary system. Their use is intended to decrease or eliminate the incidence of complications following the procedure, namely cholangitis, cholecystitis, septicemia, and pancreatitis. However, there were a few reports concerning the dosage, duration and adopting antibiotics most suitable for this purpose. The aim of this prospective comparative study is to compare the occurrence rate of post-procedural complications, such as cholangitis, bacteremia and septicemia between intravenous moxifloxacin and ceftriaxone for the prophylactic use in patients with bile duct obstruction who will undergo therapeutic ERCP procedure.

Methods: In this prospective study, a total of 160 patients (calculated by IBM SPSS Sample Power, version 3.0) with bile duct obstruction due to variable causes (bile duct stones, benign or malignant stricture, etc) will be enrolled and randomly allocated to intravenous moxifloxacin and ceftriaxone group, respectively (using simple randomization program). Intravenous moxifloxacin (400 mg/day, infused more than 60 min) or ceftriaxone (2 g/day, diluted in 40 cc of 5% dextrose water, infused more than 30 min) will be given 90 minutes before ERCP procedure, and will be given to a patient for more than 3 days if the patient develops symptoms and signs of cholangitis or septicemia.

ELIGIBILITY:
Inclusion Criteria:

* patients with bile duct obstruction due to variable causes (bile duct stones, benign or malignant stricture, etc)

Exclusion Criteria:

* pregnancy
* hypersensitivity to moxifloxacin and/or ceftriaxone
* previous antibiotic exposure or theophyllin derivatives medication within 14 days of admission
* previous history of epilepsy
* previous history of endocarditis of valvular heart disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
cholangitis | 3 days
  To compare the occurrence rate of cholangitis between the intravenous moxifloxacin and ceftriaxone group

SECONDARY OUTCOMES:
30 day mortality | 30 days
  To compare the occurrence rate of 30-day mortality between moxifloxacin and ceftriaxone treated group

CONTACTS AND LOCATIONS:
Overall Officials: Hong Joo Kim, MD, Principal Investigator — Sungkyunkwan University Kangbuk Samsung Hospital
Locations (1):
- Sungkyunkwan University Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No